CLINICAL TRIAL: NCT03925441
Title: Post-Marketing Surveillance Study of Adalimumab (Humira) for Pediatric Chronic Severe Plaque Psoriasis Patients According to the Standard for "Re-Examination of New Drugs"
Brief Title: Post-Marketing Surveillance Study of Adalimumab in Pediatric Chronic Severe Plaque Psoriasis Patients in Korea
Acronym: ped PsO rPMS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P18-839
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Psoriasis
Keywords: Post-marketing; Adalimumab; Humira; Pediatric; Chronic severe plaque psoriasis; Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric participants with chronic severe plaque psoriasis: Participants with chronic severe plaque psoriasis receiving adalimumab in routine clinical practice

SUMMARY:
The objective of this study is to evaluate the real world safety and effectiveness of adalimumab (Humira) for the treatment of Korean patients with pediatric chronic severe plaque psoriasis under a routine treatment practice.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents who are diagnosed with pediatric chronic severe plaque psoriasis.
* Prior to participating in the study, adalimumab treatment was determined according to clinical judgement of the physician.
* Participants (or legal representative) who voluntarily agreed to participate in this study and signed informed consent.

Exclusion Criteria:

* Participants with contraindication to adalimumab as listed in the approved Korean label.
* Participants with prior treatment with adalimumab.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric participants with chronic severe plaque psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Reported Any Treatment Emergent Serious Adverse Events (TESAE) OR Drug Reactions | Day 0 (informed consent) to up to 70 days following the last administration of Humira
  An adverse event (AE) is defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relations. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Percentage of Participants Who Reported Any Unexpected Treatment Emergent Adverse Events OR Drug Reactions | Day 0 (informed consent) to up to 70 days following the last administration of Humira
  An adverse event (AE) is defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relations. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. Treatment-emergent events (TEAEs) are defined as any event that began or worsened in severity after the first dose of study drug. Unexpected adverse events are the ones that do not appear on the label of the drug.

SECONDARY OUTCOMES:
Percentage of Participants Who Reported Any Treatment Emergent Non-Serious Adverse Event OR Drug Reaction | Day 0 (informed consent) to up to 70 days following the last administration of Humira
  An adverse event (AE) is defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relations. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. Treatment-emergent events (TEAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 75 From Baseline | Up to approximately 40 days
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-75 responders are the participants who achieved at least a 75% reduction (improvement) from baseline in PASI score.
Percentage of Participants Achieving PASI 90 From Baseline | Up to approximately 40 days
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-90 responders are the participants who achieved at least a 90% reduction (improvement) from baseline in PASI score.
Percentage of Participants Achieving PASI 100 From Baseline | Up to approximately 40 days
  PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). PASI-100 responders are the participants who achieved at least a 100% reduction (improvement) from baseline in PASI score.
Change in Body Surface Area (BSA) from Baseline | Up to approximately 40 days
  BSA affected by psoriasis is assessed by the Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (1):
- Ajou University Hospital /ID# 207843, Suwon, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P18-839.pdf